CLINICAL TRIAL: NCT06887920
Title: MultifocAL COntact Lenses for Myopia and Their Effect on Axial Length Elongation in Children
Brief Title: Comparison of MiSight 1-Day and Acuvue Oasys for Presbyopia in Myopic Children
Acronym: MALCOLM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pauline Kang (Other)
Collaborators: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Pauline Kang, Associate Professor, The University of New South Wales
Organization: The University of New South Wales (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC200052
Record Dates: First submitted 2025-03-14; First posted 2025-03-21 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Myopia Progressing

STUDY DESIGN:
Intervention Model Description: Non-inferiority, contralateral eye, randomised controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Acuvue Oasys for Presbyopia in the RIGHT eye (Other): Acuvue Oasys for Presbyopia in the RIGHT eye and MiSight 1-Day contact lens in the LEFT eye RIGHT eye has intervention, LEFT eye has active comparator
  Interventions: Device: Acuvue Oasys for Presbyopia
- MiSight 1-Day in the RIGHT eye (Other): MiSight 1-Day contact lens in the RIGHT eye and Acuvue Oasys for Presbyopia in the LEFT eye RIGHT eye has active comparator, LEFT eye has intervention
  Interventions: Device: MiSight 1 Day

INTERVENTIONS:
Device: Acuvue Oasys for Presbyopia — ACUVUE OASYS for PRESBYOPIA contact lenses will be prescribed to children with myopia to be worn in one eye for 10 hours a day for one year.
  Arms: Acuvue Oasys for Presbyopia in the RIGHT eye
Device: MiSight 1 Day — MiSight 1 Day contact lenses will be prescribed to children with myopia to be worn in one eye for 10 hours a day for one year.
  Arms: MiSight 1-Day in the RIGHT eye

SUMMARY:
This study will compare the effects on myopia progression over the course of one year for eyes wearing MiSight 1 Day contact lenses compared to ACUVUE OASYS for PRESBYOPIA contact lenses.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6-12 years (inclusive)
2. Is willing to wear soft contact lenses daily
3. Spherical equivalent myopic refractive error between -0.50 to -5.00 D in each eye and astigmatism < 1.00 D
4. Best corrected logMAR visual acuity of 0.1 or better in both eyes
5. Good ocular and general health
6. No previous use of myopia control interventions for more than 1 month or within the last 30 days
7. Competent enough in English to be able to fully understand the participant information and consent form

Exclusion Criteria:

1. Strabismus at distance or near, amblyopia or significant anisometropia (>1D)
2. Systemic or ocular conditions that may affect contact lens use (e.g., allergy) or that may affect refractive development (e.g., ptosis)
3. Previous history of ocular surgery, trauma, or chronic ocular disease
4. Contraindications to contact lens use
5. Ocular or systemic medication use which may interfere or interact with contact lens wear or ocular development
6. Plans to migrate or move during the study
7. Child, parents or guardians not willing to comply with treatment and/or follow-up schedule

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Axial length progression | 1 month, 6 months and 12-months post intervention commencement. Initial protocol also included 3-month time point, but the 3-month visit was updated to a telehealth consultation due to COVID-19 restrictions. Updated after 9 participants.
  Change in Axial Length between two eyes measured by laser interferometry (IOL Master)
Cycloplegic autorefraction | 1 month, 6 months and 12-months post intervention commencement. Initial protocol also included 3-month time point, but the 3-month visit was updated to a telehealth consultation due to COVID-19 restrictions. Updated after 9 participants.
  Change in Autorefraction between two eyes as measured by autorefractor

SECONDARY OUTCOMES:
Subjective refraction | 1 month, 6 months and 12-months post intervention commencement. Initial protocol also included 3-month time point, but the 3-month visit was updated to a telehealth consultation due to COVID-19 restrictions. Updated after 9 participants.
  Change in subjective refraction between two eyes using phoropter or trial frame
Estimates of outdoor time and near work | 1-month, 6-month and 12-month study visits. Also 3-month and 9-month telehealth visits. 3-month visit was changed to telehealth and 9-month visit added after already enrolling 9 participants.
  Estimates of time spent outdoors and on near work with study specific questionnaire. Duration will be reported in minutes or hours.
Quality of Life (PREP2) | Baseline, 6-month and 12-month study visits. Added after already enrolling 9 participants.
  Quality of Life measured using the PREP2 survey. Scores are derived from a scale between 0 to 100, with higher values incating better Quality of Life.
Quality of Life (PedEyeQ) | Baseline, 6-month and 12-month study visits. Added after already enrolling 9 participants.
  Quality of Life measured using the PedEyeQ survey. Scores are derived from a scale between 0 to 100, with higher values incating better Quality of Life.
Treatment adherence (Questions) | 1-month, 6-month and 12-month study visits. Added to initial protocol prior to enrolment commencement.
  Contact lens wear duration will be calculated from study-specific questionnaire conducted at study visits. Duration will be reported as hours per day and days per week.
Treatment adherence (Text-message surveys) | Study month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12. 1-month, 6-month and 12-month study visits. Added to initial protocol prior to enrolment commencement.
  Contact lens wear duration will be calculated from study-specific questionnaire sent via text-message. Duration will be reported as hours per day and days per week.

OTHER OUTCOMES:
Corneal topography | 1 month, 6 months and 12-months post intervention commencement. Initial protocol also included 3-month time point, but the 3-month visit was updated to a telehealth consultation due to COVID-19 restrictions. Updated after 9 participants.
  Change in Corneal topography measurements between two eyes as measured by corneal topographer (Oculus Keratograph, Medmont E300)
Amplitude of Accommodation | 1 month, 6 months and 12-months post intervention commencement. Initial protocol also included 3-month time point, but the 3-month visit was updated to a telehealth consultation due to COVID-19 restrictions. Updated after 9 participants.
  Change in amplitude of accommodation between the two eyes with push up test
Visual acuity | 1 month, 6 months and 12-months post intervention commencement. Initial protocol also included 3-month time point, but the 3-month visit was updated to a telehealth consultation due to COVID-19 restrictions. Updated after 9 participants.
  Change in distance and near vision between the two eyes using visual acuity charts
Anterior Chamber Depth | 1 month, 6 months and 12-months post intervention commencement. Initial protocol also included 3-month time point, but the 3-month visit was updated to a telehealth consultation due to COVID-19 restrictions. Updated after 9 participants.
  Change in anterior chamber depth between the two eyes with laser interferometry (IOL Master) and optical coherence tomography (Casia SS-1000)
Corneal radii | 1 month, 6 months and 12-months post intervention commencement. Initial protocol also included 3-month time point, but the 3-month visit was updated to a telehealth consultation due to COVID-19 restrictions. Updated after 9 participants.
  Change in corneal radii between the two eyes with laser interferometry (IOL Master).
Lens thickness | 1 month, 6 months and 12-months post intervention commencement. Initial protocol also included 3-month time point, but the 3-month visit was updated to a telehealth consultation due to COVID-19 restrictions. Updated after 9 participants.
  Change in lens thickness between the two eyes with laser interferometry (IOL Master).
Posterior segment depth | 1 month, 6 months and 12-months post intervention commencement. Initial protocol also included 3-month time point, but the 3-month visit was updated to a telehealth consultation due to COVID-19 restrictions. Updated after 9 participants.
  Change in posterior segment depth measurements with optical coherence tomography
Pupils | 1 month, 6 months and 12-months post intervention commencement. Initial protocol also included 3-month time point, but the 3-month visit was updated to a telehealth consultation due to COVID-19 restrictions. Updated after 9 participants.
  Change in pupillary measurements as measured by pupillometer

CONTACTS AND LOCATIONS:
Locations (1):
- University of New South Wales, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dang R, Hui A, Jalbert I, Kho D, Vi M, Briggs N, Kang P. MultifocAL COntact Lenses for Myopia (MALCOLM) control in Australian children: a study protocol for a double-blind, contralateral eye, non-inferiority, randomised controlled clinical trial. BMJ Open. 2025 Apr 14;15(4):e086173. doi: 10.1136/bmjopen-2024-086173. PMID 40228855